CLINICAL TRIAL: NCT05578313
Title: Inflammatory Bowel Diseases (IBD) Cannabis Registry
Acronym: IBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eli Sprecher, MD (Other Government)
Responsible Party: Sponsor-Investigator, Eli Sprecher, MD, PI, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TLV_0276-19
Record Dates: First submitted 2021-06-30; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease; Ulcerative Colitis; Pouchitis; Healthy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Pouchitis | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Baseline and follow up study visits will include biologic samples collection (blood, feces) from which blood levels of complete blood count (CBC), Albumin, Liver enzymes (ALT, AST, ALP), lipid panel (Total cholesterol, LDL, HDL, triglycerides), creatinine, fasting glucose, C-reactive protein (CRP), drug levels and antibodies (for patients treated with thiopurines and biologics), and fecal levels of Calprotectin will be measured.
  White blood cells will be separated and stored for mRNA analysis of cannabinoid metabolism. Only RNA fractions will be extracted and analyzed, no DNA will be assessed and no genetic sequencing will be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- • Group 1 (study group): IBD patients prescribed cannabis as treatment of their bowel disease.
  Interventions: Drug: Medical Cannabis
- • Group 2 (Control group): One hundred healthy patients who do not use cannabis and are not eligible or not interested to commence this intervention.
- • Group 3 (control group): Up to 100 IBD patient who experience pain and do not use cannabis
- • Group 4 (control group): Up to 100 IBD patient who do not experience pain and do not use cannabis
- • Group 5 (Cannabis responders group): up to 100 IBD patients previously prescribed cannabis and were identified to have positive effect on their disease

INTERVENTIONS:
Drug: Medical Cannabis — Patients will be observed throughout their treatment with medical cannabis, prescribed to them by for clinically treating their disease (treatment is not an intervention of the study).
  Groups: • Group 1 (study group)

SUMMARY:
The inflammatory bowel diseases (IBDs), ulcerative colitis (UC) and Crohn's disease (CD), are characterized by lifelong relapsing-remitting gastrointestinal inflammation, with symptoms of abdominal pain, diarrhea, and rectal bleeding during active disease. Medical therapy reduces intestinal inflammation and ameliorates symptoms. Medical cannabis has recently been added to the arsenal of symptom-reducing measures in IBD. Though the efficacy of THC and CBD have been established as the two most dominant ingredients of cannabis, the rest of the plant phytochemicals are unknown, and effects on patients are not yet determined.

DETAILED DESCRIPTION:
Hypothesis (es) and Aims:

Prospectively follow IBD patients receiving medical cannabis as treatment of their disease (group 1) in comparison to the following control groups:

2) Healthy patients who do not use cannabis; 3) IBD patients who experience pain and do not use cannabis; 4) IBD patients who do not experience pain and do not use cannabis; 5) IBD patients previously prescribed cannabis and were identified to have positive effect on their disease

• Specific aims: a prospective trial to determine whether cannabis can induce remission in patients with IBD.

* To identify treatment regimens associated with treatment success in IBD patients.
* To identify treatment regimens associated with treatment side effects in IBD patients.
* To analyze the optimal drug level for disease management in various IBD patient types.

  * Study design:

    * A prospective cohort study
    * Setting: prospectively collect clinical, behavioral, dietary and environmental data of IBD patients receiving medical cannabis as treatment of their disease. Data will be collected according to a uniform standardized protocol specifically adapted to the needs of the study.
  * Study population:

Eligible IBD patients treated at the IBD clinic in the Tel Aviv Medical Center participating in the study, which have signed an informed consent form and answered to all the study inclusion criteria. Patients will be informed of the study by their treating physician, recruited and followed throughout the follow-up period by study coordinators.

This study will include five patient groups:

* Group 1 (study group): IBD patients prescribed cannabis as treatment for their bowel disease.
* Group 2 (Control group): One hundred healthy patients who do not use cannabis and are not eligible or not interested to commence this intervention.
* Group 3 (control group): Up to 100 IBD patient who experience pain and do not use cannabis
* Group 4 (control group): Up to 100 IBD patient who do not experience pain and do not use cannabis
* Group 5 (Cannabis responders group): up to 100 IBD patients previously prescribed cannabis and were identified to have positive effect on their disease

  *Study plan:
* Among the study group :

At baseline, demographic characteristics, medical history, concomitant medication assessment, disease related therapy and failed therapy will be documented.

Study visits:

Among the study group: recruitment at time 0, after one month (±14 days) of treatment, at three months (±21 days) and at 6 months (±30 days) of therapy (end of study), will be conducted, in which patients will be asked to fill in questionnaires, give biologic samples, undergo clinical, anthropometric and nutritional evaluation and physician assessment and monitoring of therapy, safety and adverse events. The cannabis producing company, composition, quantity and way of consumption will be documented.

•Among control group and Cannabis responders group: Healthy controls will be samples once at baseline. All IBD control groups (groups 3-5) will be followed up similarly as the study group and will undergo all sampling and questionnaires, at times 0, 3, 6 months (excluding the 1 month cannabis dose adjustment meeting).

Patients will be asked to inform in case of relapse during the follow up period and provide stool and blood samples before therapy is changed. At relapse time point, disease activity index will be recorded and questionnaires will be completed.

*Sample collection: Baseline and follow up study visits will include biologic samples collection (blood, feces) from which blood levels of complete blood count (CBC), Albumin, Liver enzymes (ALT, AST, ALP), lipid panel (Total cholesterol, LDL, HDL, triglycerides), creatinine, fasting glucose, C-reactive protein (CRP), drug levels and antibodies (for patients treated with thiopurines and biologics), and fecal levels of Calprotectin will be measured.

White blood cells will be separated and stored for m RNA analysis of cannabinoid metabolism. Only RNA fractions will be extracted and analyzed, no DNA will be assessed and no genetic sequencing will be performed . In addition, 10 ml of blood will be drawn for analysis of Th17 cells. CD4 T cells will be purified from peripheral blood of IBD patients by RosetteSep™ Human CD4+ T Cell Enrichment Cocktail kit. STAT3 and IL-17 levels will be analyzed. The samples analysis will be done at Dedi Meiri's lab at the Technion-IIT. Serum, and fecal samples will be stored at -80◦C for future analysis after being authorized by the IRB and by law including cannabis phytochemical analysis (10ml of each) on WBC and on biopsies when available and for fecal microbiome analysis. In appendix A- a detailed list of all tests in each visit.

*Endoscopic evaluation: In patients who will undergo a standard of care endoscopic examination for clinical reasons: these will include mucosal and histologic assessment for disease severity (SES-CD and MAYO score for CD and UC patients respectively, PDAI for Pouchitis patients).

Mucosal biopsies will be collected from inflamed and healthy areas, and from standard areas of the GI track (table 1), sent for histology assessment and stored for future analysis after being authorized by the IRB and by law. These samples will be stored in RNA Later snapped frozen and stored at -80◦c until analysis. No more than 10 samples will be collected during endoscopy including samples for clinical assessment. Samples from recto-sigmoid junction (20 cm from anus) will be taken in every colonoscopy, regardless of the status of inflammation.

*Biologic sample handling: Samples will be stored at -80◦c while coded with no identifying information; access to samples will be restricted to the study staff only. Samples will be stored up to 10 years from final data collection.

In this study, serum and fecal samples analyzed will include those gathered from protocol number 0276-19 and from protocol number 0250-17 in patients using medical cannabis only. In the later group, samples will be used only if the patient had agreed for use of samples in other studies other than 0250-17. To both studies, Professor Nitsan Maharshak is PI.

*Questionnaires:

Baseline and follow up study visits will include data collection from the following:

* Documentation of cannabis therapy: consumption method, quantity, THC/CBD concentration and cannabis strain/ barcode of preparation
* Food frequency questionnaire
* Food diary from last 3 days
* Lifestyle questionnaire
* Medical management questionnaire (IBD SES- self efficacy scale questionnaire)
* Patient reported outcomes (PROMIS) questionnaires
* Medical cannabis treatment evaluation questionnaire and Adverse events
* Big Five personality traits

Anthropometric and nutritional evaluation:

* Patients weight (kg), height (m), waist circumference (cm) will be documented at each study visit, and body mass index (BMI) will be calculated.
* Nutritional status will be evaluated by a MUST questionnaire

  *Study endpoints: the study will follow patients throughout 6 months of treatment and follow disease remission (clinical/biochemical) or exacerbation.
* Disease remission:

  * Reduction in appropriate clinical scores
  * Decrease in serum CRP or fecal CLP
  * Endoscopic remission
* Disease exacerbation:

  * Increase in appropriate clinical score
  * Increase in fecal calprotectin levels (>250mg/gr OR 100 units higher than baseline levels)
  * Emergency room visit due to disease symptoms, hospitalization, non-elective surgery.
  * Diagnosis of active disease by endoscopy or imaging
  * Medical treatment change by treating physician

    * Statistical analysis:

Statistical analyses will be performed using SPSS version 23.0 for Windows. Patients who adhere to the study's protocol (defined as preforming ≥ 80% of exercises) will be included in data analysis. An intention-to-treat analysis will include patients excluded because of non-adherence to the intervention.

Descriptive statistics will be used to describe the distribution of variables associated with characteristics of the study sample. Continuous variables will be presented as means± SD and dichotomous/categorical variables as proportions. The normality of the distribution of continuous variables will be tested by the Kolmogorov-Smirnov test. If normality is rejected, non-parametric tests will be used.

Univariate analysis: To test the association between continuous variables with normal distribution, the Pearson correlation coefficient will be performed. To test associations between continuous variables which do not distribute normally or for ordinal variable, the spearman correlation coefficient will be used. To test differences in continuous variables between the treatments arms the t-test for independent groups (or Mann-Whitney test for non-normally distributed variables) will be performed. For comparison of dichotomous or categorical variables the Chi-square test will be performed.

To compare baseline to end of treatment parameters within arms for continuous variables the t-test for dependent groups will be performed (or Wilcoxson test for non-normally distributed variables), in dichotomous/categorical variables the McNemar Test will be performed.

To test differences in continuous variables between the treatment groups in numbers of time points the Mix model for repeated measures will be performed. To test differences in dichotomous/categorical variables between the treatment groups in numbers of time points Generalized estimating equation will be performed.

ELIGIBILITY:
Inclusion Criteria:

Patients (male and female, age 18-80 years) diagnosed with Crohn's disease (CD), ulcerative colitis (UC) or pouchitis, and healthy volunteers.

All patients will sign an informed consent form. IBD patients who are recruited to group 3 will be included if they report mild-severe abdominal pain in clinical questioning of clinical activity (Harvey-Bradshaw index).

Healthy participants recruited to group 2 will be healthy volunteers with no prior/current use of medical cannabis

Exclusion Criteria:

* Inability to sign an informed consent and complete the study protocol
* Unstable or uncontrolled medical disorder, or severe systemic disease (other than IBD)
* Participating in clinical interventional trial unrelated to cannabis derived preparations
* Ileostomy/ colostomy
* Pregnancy or intent to become pregnant in the next 6 month or breast feeding during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population:
  Eligible IBD patients treated at the IBD clinic in the Tel Aviv Medical Center participating in the study, which have signed an informed consent form and answered to all the study inclusion criteria. Patients will be informed of the study by their treating physician, recruited and followed throughout the follow-up period by study co-ordinators.
  This study will include five patient groups:
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2023-07-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Determine patients clinical response rates using Harvey-Bradshaw Index (HBI) in Crohn's disease patients receiving cannabis at week 4 | week 4
  Disease clinical response will be measured as the change in HBI scores from baseline to week 4.
  A clinical response is defined as reduction of at least 3 points in HBI score, ∆HBI>3 in patients with baseline HBI>7.
  Harvey-Bradshaw Index (HBI) is a tool for assessing the degree of illness (activity) in patient's with Crohn's disease. Higher score means higher disease activity and severity. A drop > 3 is considered a clinical response.
Determine the clinical response rates using SCCAI (Simple Clinical Colitis Activity Index) in patients with Ulcerative Colitis receiving cannabis at week 4 | week 4
  Disease clinical response will be measured as the change in SCCAI scores from baseline to week 4.
  A clinical response is defined as reduction of at list 30% in SCCAI score, ∆SCCAI>30% for Ulcerative Colitis
  SCCAI (Simple Clinical Colitis Activity Index) is used to assess the severity of symptoms in people who suffer from ulcerative colitis. Score range from 0 to 19 points 0<SCCAI<19. Higher score means higher disease activity and severity.
Determine patients clinical response rates using Harvey-Bradshaw Index (HBI) in Crohn's disease patients receiving cannabis at week 12 | week 12
  Disease clinical response will be measured as the change in HBI scores from baseline to week 12.
  A clinical response is defined as reduction of at least 3 points in HBI score, ∆HBI>3 in patients with baseline HBI>7.
  Harvey-Bradshaw Index (HBI) is a tool for assessing the degree of illness (activity) in patient's with Crohn's disease. Higher score means higher disease activity and severity. A drop > 3 is considered a clinical response.
Determine the clinical response rates using SCCAI (Simple Clinical Colitis Activity Index) in patients with Ulcerative Colitis receiving cannabis at week 12 | week 12
  Disease clinical response will be measured as the change in SCCAI scores from baseline to week 12.
  A clinical response is defined as reduction of at list 30% in SCCAI score, ∆SCCAI>30% for Ulcerative Colitis
  SCCAI (Simple Clinical Colitis Activity Index) is used to assess the severity of symptoms in people who suffer from ulcerative colitis. Score range from 0 to 19 points 0<SCCAI<19. Higher score means higher disease activity and severity.
Determine patients clinical response rates using Harvey-Bradshaw Index (HBI) in Crohn's disease patients receiving cannabis at week 24 | Week 24
  Disease clinical response will be measured as the change in HBI scores from baseline to week 24.
  A clinical response is defined as reduction of at least 3 points in HBI score, ∆HBI>3 in patients with baseline HBI>7.
  Harvey-Bradshaw Index (HBI) is a tool for assessing the degree of illness (activity) in patient's with Crohn's disease. Higher score means higher disease activity and severity. A drop > 3 is considered a clinical response.
Determine the clinical response rates using SCCAI (Simple Clinical Colitis Activity Index) in patients with Ulcerative Colitis receiving cannabis at week 24 | Week 24
  Disease clinical response will be measured as the change in SCCAI scores from baseline to week 24.
  A clinical response is defined as reduction of at list 30% in SCCAI score, ∆SCCAI>30% for Ulcerative Colitis
  SCCAI (Simple Clinical Colitis Activity Index) is used to assess the severity of symptoms in people who suffer from ulcerative colitis. Score range from 0 to 19 points 0<SCCAI<19. Higher score means higher disease activity and severity.

SECONDARY OUTCOMES:
Determine clinical remission rates using Harvey-Bradshaw Index (HBI) in Crohn's disease patients receiving cannabis at weeks 4 | week 4
  Disease remission will be defined by HBI <5
  Higher HBI clinical score means higher disease severity:
  Remission<5 Mild Disease 5-7 Moderate Disease 8-16 Severe Disease >16
Determine clinical remission rates using SCCAI (Simple Clinical Colitis Activity Index) in patients with Ulcerative Colitis receiving cannabis at week 4 | week 4
  Disease remission will be defined by SCCAI <3
  SCCAI (Simple Clinical Colitis Activity Index) score range from 0 to 19. Higher score means higher disease severity.
Determine clinical remission rates using Harvey-Bradshaw Index (HBI) in Crohn's disease patients receiving cannabis at weeks 12 | week 12
  Disease remission will be defined by HBI <5
  Higher HBI clinical score means higher disease severity:
  Remission<5 Mild Disease 5-7 Moderate Disease 8-16 Severe Disease >16
Determine clinical remission rates using SCCAI (Simple Clinical Colitis Activity Index) in patients with Ulcerative Colitis receiving cannabis at week 12 | week 12
  Disease remission will be defined by SCCAI <3
  SCCAI (Simple Clinical Colitis Activity Index) score range from 0 to 19. Higher score means higher disease severity.
Determine clinical remission rates using Harvey-Bradshaw Index (HBI) in Crohn's disease patients receiving cannabis at weeks 24 | week 24
  Disease remission will be defined by HBI <5
  Higher HBI clinical score means higher disease severity:
  Remission<5 Mild Disease 5-7 Moderate Disease 8-16 Severe Disease >16
Determine clinical remission rates SCCAI (Simple Clinical Colitis Activity Index) in patients with Ulcerative Colitis receiving cannabis at week 24 | week 24
  Disease remission will be defined by SCCAI <3
  SCCAI (Simple Clinical Colitis Activity Index) score range from 0 to 19. Higher score means higher disease severity.
Determine endoscopic response rates using Simple Endoscopic Score for Crohn Disease (SES-CD) in patients with Crohn's disease receiving cannabis at weeks 4 | week 4
  Endoscopic response will be defined as decrease of ≥50% in SES-CD score from baseline to week 4
  Higher SES-CD score means higher disease activity and severity. A drop > 50% is considered an endoscopic response
Determine endoscopic response rates using Mayo score in patients with Ulcerative Colitis receiving cannabis at weeks 4 | week 4
  Endoscopic response will be defined as reduction in Endoscopic Mayo score ≤ 1 for Ulcerative Colitis
  Endoscopic Mayo score range from 0-3. Higher score means higher disease severity
Determine endoscopic response rates using Simple Endoscopic Score for Crohn Disease (SES-CD) in patients with Crohn's disease receiving cannabis at weeks 12 | week 12
  Endoscopic response will be defined as decrease of ≥50% in SES-CD score from baseline to week 12
  Higher SES-CD score means higher disease activity and severity. A drop > 50% is considered an endoscopic response
Determine endoscopic response rates using Mayo score in patients with Ulcerative Colitis receiving cannabis at weeks 12 | week 12
  Endoscopic response will be defined as reduction in Endoscopic Mayo score ≤ 1 for from baseline to week 12
  Endoscopic Mayo score range from 0-3. Higher score means higher disease severity
Determine endoscopic response rates using Simple Endoscopic Score for Crohn's Disease (SES-CD) in patients with Crohn's disease receiving cannabis at weeks 24 | week 24
  Endoscopic response will be defined as decrease of ≥50% in SES-CD score from baseline to week 24
  Higher SES-CD score means higher disease activity and severity. A drop > 50% is considered an endoscopic response
Determine endoscopic response rates using Mayo score in patients with Ulcerative Colitis receiving cannabis at weeks 24 | week 24
  Endoscopic response will be defined as reduction in Endoscopic Mayo score ≤ 1 for from baseline to week 24
  Endoscopic Mayo score range from 0-3. Higher score means higher disease severity
Determine endoscopic remission rates using Simple Endoscopic Score for Crohn's Disease (SES-CD) in patients with Crohn's disease receiving cannabis at week 4 | week 4
  Endoscopic remission will be defined as SES-CD<4 for Crohn's disease
  SES-CD ranges from a minimum score o and has no high limit. Higher SES-CD score means higher disease severity and activity.
Determine endoscopic remission rates using Mayo score in patients with Ulcerative Colitis receiving cannabis at weeks 4 | week 4
  Endoscopic remission will be defined as Endoscopic Mayo score = 0 for ulcerative colitis
  Endoscopic Mayo score range from 0-3. Higher score means higher disease severity
Determine endoscopic remission rates using Simple Endoscopic Score for Crohn's Disease (SES-CD) in patients with Crohn's disease receiving cannabis at week 12 | week 12
  Endoscopic remission will be defined as SES-CD<4 for Crohn's disease
  SES-CD ranges from a minimum score o and has no high limit. Higher SES-CD score means higher disease severity and activity.
Determine endoscopic remission rates using Mayo score in patients with Ulcerative Colitis receiving cannabis at weeks 12 | week 12
  Endoscopic remission will be defined as Endoscopic Mayo score = 0 for ulcerative colitis
  Endoscopic Mayo score range from 0-3. Higher score means higher disease severity
Determine endoscopic remission rates using Simple Endoscopic Score for Crohn's Disease (SES-CD) in patients with Crohn's disease receiving cannabis at week 24 | week 24
  Endoscopic remission will be defined as SES-CD<4 for Crohn's disease
  SES-CD ranges from a minimum score o and has no high limit. Higher SES-CD score means higher disease severity and activity.
Determine endoscopic remission rates using Mayo score in patients with Ulcerative Colitis receiving cannabis at weeks 24 | week 24
  Endoscopic remission will be defined as Endoscopic Mayo score = 0 for Ulcerative Colitis
  Endoscopic Mayo score range from 0-3. Higher score means higher disease severity

OTHER OUTCOMES:
Assess the effect of cannabis treatment on pain levels using visual analog scale (VAS) in patients with IBD, after 1 month of treatment | week 4
  Pain levels will be measured using pain visual analog scale (VAS)
  VAS scale range from 0 to 10, where 0 means no pain and higher score means worse pain
Assess the effect of cannabis treatment on pain levels using visual analog scale (VAS) in patients with IBD, after 3 month of treatment | week 12
  Pain levels will be measured using pain visual analog scale (VAS)
  VAS scale range from 0 to 10, where 0 means no pain and higher score means worse pain
Assess the effect of cannabis treatment on pain levels using visual analog scale (VAS) in patients with IBD, after 6 month of treatment | week 24
  Pain levels will be measured using pain visual analog scale (VAS)
  VAS scale range from 0 to 10, where 0 means no pain and higher score means worse pain
Assess the effect of cannabis treatment on sleep quality using the Pittsburgh Sleep Quality Index (PSQI) in patients with IBD after 1 month of treatment | week 4
  Sleep quality will be measured using the PSQI
  PSQI has a range of 0-21; higher score indicate worse sleep quality.
Assess the effect of cannabis treatment on sleep quality using the Pittsburgh Sleep Quality Index (PSQI) in patients with IBD after 3 month of treatment | week 12
  Sleep quality will be measured using the PSQI
  PSQI has a range of 0-21; higher score indicate worse sleep quality.
Assess the effect of cannabis treatment on sleep quality using the Pittsburgh Sleep Quality Index (PSQI) in patients with IBD after 6 month of treatment | week 24
  Sleep quality will be measured using the PSQI
  PSQI has a range of 0-21; higher score indicate worse sleep quality.
Assess the safety of cannabis treatment in patients with IBD after 1 month of treatment | 4 weeks
  The safety of cannabis treatment will be measured using Common Terminology Criteria for Adverse Events (CTCAE)
Assess the safety of cannabis treatment in patients with IBD after 3 month of treatment | 12 weeks
  The safety of cannabis treatment will be measured using Common Terminology Criteria for Adverse Events (CTCAE)
Assess the safety of cannabis treatment in patients with IBD after 6 month of treatment | 24 weeks
  The safety of cannabis treatment will be measured using Common Terminology Criteria for Adverse Events (CTCAE)
Assess the effect of cannabis treatment on quality of life using medical management questionnaire (IBD self-efficacy scale) in patients with IBD | week 24
  Quality of life will be measured using IBD self-efficacy scale questionnaire
  The overall score of the IBD-SES ranges from 29 to 290 with a lower score indicating lower SE.
Assess the effect of cannabis treatment on quality of life Patient Reported Outcomes (PROMIS) questionnaire in patients with IBD | week 24
  Quality of life will be measured using Patient Reported Outcomes (PROMIS) questionnaire
  PROMIS measures use T-scores. A higher PROMIS T-score represents more of the concept being measured (negative or positive)
Assess personality traits of patients with IBD favoring cannabis treatment using the Big Five personality traits questionnaire | week 24
  Personality traits will be measured using the Big Five personality traits questionnaire
  Each personality type will have a score between 0-40. Higher scores equal stronger personality type.

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel